CLINICAL TRIAL: NCT03450369
Title: A Phase 1B Dose Escalating Study of the Safety, Short-Term Engraftment and Action of a Singly-Applied NB01 in Adults With Moderate Acne
Brief Title: A Study of the Safety, Engraftment, and Action of NB01 in Adults With Moderate Acne
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Naked Biome, Inc. (Industry)
Collaborators: Dermatology Research Institute (Other); QST Consultations, Ltd. (Industry); Science 37 (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NB01-P1BSA
Record Dates: First submitted 2018-02-13; First posted 2018-03-01 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: Open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NB01 (Experimental): NB01 is a live probiotic containing a single strain of P. acnes, frozen, on a pad, in a single use pouch, for topical application.
  Open label and dose escalation of a single application of NB01 to subjects with moderate acne, with approximately 5 subjects assigned to lower bound dose before escalation to upper bound dose.
  Interventions: Biological: NB01

INTERVENTIONS:
Biological: NB01 — Use an existing therapy designed to kill existing facial bacterial followed by populating facial skin with a single application of NB01

SUMMARY:
Acne vulgaris is a multifactorial disease caused by overgrowth of Propionibacterium acnes (P. acnes), impaction of hair follicles, excessive sebum production and hormonal dysregulation. Recent literature from the Human Microbiome Project has shown there are unique microbial signatures specific to healthy and acne disease states.

From this data, the investigators hypothesize that by eliminating resident disease-associated bacterial strains and replacing them with health-associated strains, recurrences/fares of acne may be improved, mitigated, and prevented. Instead of current approaches which focus on eliminating all bacteria from the skin, the investigators aim to deliver healthy bacteria to restore the skin to a healthy state via this replacement therapy.

The investigators aim to test this in a Phase Ib single application study evaluating the safety, tolerability, and clinical impact that a single application of NB01, a live strain of P. acnes, has on adult subjects with moderate acne.

DETAILED DESCRIPTION:
A Phase 1B Dose Escalating Study of the Safety, Short-Term Engraftment and Action of a Singly Applied NB01 in Adults with Moderate Acne

Acne vulgaris is a multifactorial disease caused by overgrowth of Propionibacterium acnes (P. acnes), impaction of hair follicles, excessive sebum production and hormonal dysregulation. Recent literature from the Human Microbiome Project has shown there are unique microbial signatures specific to healthy and acne disease states.

From this data, the investigators hypothesize that by eliminating resident disease-associated bacterial strains and replacing them with health-associated strains, recurrences/fares of acne may be improved, mitigated, and prevented. Instead of current approaches which focus on eliminating all bacteria from the skin, the investigators aim to deliver healthy bacteria to restore the skin to a healthy state via this replacement therapy.

The investigators aim to test this in a Phase Ib single application study evaluating the safety, tolerability, and clinical impact that a single application of NB01 has on adult subjects with moderate acne. Investigators will be profiling the change in microbiome over the course of therapy to determine if exogenously delivered bacteria can populate the skin (engraftment) and cause a shift in the microbiome safely and subsequently impact acne biomarkers that may correlate with clinical disease.

The investigators intend for this therapy to eventually be used in acne subjects with ages ranging from 13-40, and all disease severities as either monotherapy for mild to mild/moderate acne and as an adjuvant therapy for moderate to severe acne at all body sites, with special attention to facial involvement.

This approach is standard to acne therapy whereby mild disease will be treated with a monotherapy (i.e., topical Benzoyl peroxide [BPO]) and moderate/severe disease will be treated with various combinatory regimens (topical antibiotics, BPO, topical retinoids, oral antibiotics).

Primary Objectives:

1. To determine the safety profile and tolerability of a singly applied NB01
2. To define engraftment of a singly applied topical NB01.
3. Dose schedule determination based on engraftment

Secondary Objective: To evaluate clinical efficacy using FDA standards of acne clinical assessments, namely the Investigator Global Assessment (IGA) and acne lesion counts of a singly applied NB01.

Approximately 10 total male and female adult subjects combined with moderate, non-cyclical acne will be enrolled into the trial. Approximately five (5) subjects will be assigned to each dose schedule

This is a single topical application study of live bacteria for the study of acne in adult subjects.

Subject participation in the trial will range from 5 weeks to 2 months.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed e-consent.
2. Males and Females ages 18-40.
3. Acne severity: Moderate (Grade 3 on 5-point IGA scale and Moderate on an acne lesion count scale (Appendix B [Section 12.2], IGA and Lesion Count Acne Grading).
4. Acne treatment-free period (including topical or oral antibiotics, retinoids, laser therapy, topical dapsone, topical azelaic acid, facial peels, dermabrasion, sulfacetamide sulfur, and salicylic acid), of at least 3 weeks prior to e-consent (with the exception of BPO pre-treatment under this protocol).
5. Lesion count: A minimum of at least a total of 15 inflammatory lesions (papules plus pustules), with a minimum of 10 inflammatory lesions within the designated application area (cheek/nose).
6. Females with non-cyclical acne.
7. Females of childbearing potential willing to use adequate contraception (e.g., total abstinence, intrauterine device (IUD), barrier method with spermicide, surgical sterilization or surgically sterilized partner, Depo-Provera®, Norplant®, or NuvaRing® for the duration of the Screening Period and during study participation. All oral contraceptive and hormonal implants will need to have been initiated and on a stable dose for at least 3 months prior to the screening period. Women of childbearing potential are defined as any female who has experienced menarche and who is NOT permanently sterile or postmenopausal; postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause.
8. Male participants willing to use an acceptable method of contraception (e.g., total abstinence, barrier methods with spermicide, surgical sterilization or surgically sterilized partner) during study participation.

Exclusion Criteria:

1. Active bacterial, viral, or fungal skin infections.
2. Any noticeable breaks or cracks in the skin on the face, including severely excoriated skin or skin with open or weeping wounds suggestive of an active infection or increased susceptibility to infection.
3. Comorbid skin conditions in the area of application.
4. Active periodontal disease or ongoing procedures (e.g., gum grafting).
5. History/current ocular infections/surgeries within 6 months of enrollment, with the exception of any history of cataracts.
6. History of sarcoidosis.
7. History septic joints/endocarditis.
8. Participants with Netherton's syndrome or other genodermatoses that result in a defective epidermal barrier.
9. Sensitivity to or difficulty tolerating glycerin, polyethylene glycol.
10. History of isotretinoin use, with the exception of sub-therapeutic treatment within 8 weeks of enrollment.
11. Less than 80% compliance with BPO, or less than 5 days' worth of BPO pre-treatment (whichever is greater) during the Screening period.
12. Current major systemic comorbid conditions.
13. Currently participating in (or within 8 weeks of enrollment) another acne trial or other investigational drug.
14. Participants with prosthetic heart valves, pacemakers, intravascular catheters, or other foreign or prosthetic devices/implantable devices/hardware.
15. Participants with close contact (e.g., spouses, children, or members in the same household) with prosthetic heart valves, pacemakers, intravascular catheters, or other foreign or prosthetic devices/implantable devices/hardware.
16. Known chronic human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV) infections.
17. History of malignancy (with the exception of non-melanoma skin cancer).
18. Immunosuppression (such as resulting from transplantation, immunosuppressive therapy, active HIV infection/acquired immune deficiency syndrome [AIDS], neutropenia).
19. Major surgical procedure, open biopsy, or significant traumatic injury within 14 days of initiating study drug (unless the wound has healed), or anticipation of the need for major surgery during the study.
20. The presence of a medical or psychiatric condition, history of drug or alcohol abuse that, in the opinion of the PI, makes the subject inappropriate for study inclusion.
21. Participants with close contacts (e.g., spouses, children, or members in the same household) that have severe barrier defects or are immunocompromised.
22. Inability or unwillingness of participant to comply with study protocol procedures.
23. Pregnant or lactating females, or females who desire to become pregnant and/or breast feed within the duration of study participation.
24. Imprisonment or under legal guardianship.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Taylor, MD, Study Director — CEO
Locations (1):
- Dermatology Research Associates, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Initially there is no plan to share individual participant data (IPD). This may change later as the clinical plan develops.

REFERENCES:
- [Background] Achermann Y, Goldstein EJ, Coenye T, Shirtliff ME. Propionibacterium acnes: from commensal to opportunistic biofilm-associated implant pathogen. Clin Microbiol Rev. 2014 Jul;27(3):419-40. doi: 10.1128/CMR.00092-13. PMID 24982315
- [Background] Akaza N, Akamatsu H, Numata S, Yamada S, Yagami A, Nakata S, Matsunaga K. Microorganisms inhabiting follicular contents of facial acne are not only Propionibacterium but also Malassezia spp. J Dermatol. 2016 Aug;43(8):906-11. doi: 10.1111/1346-8138.13245. Epub 2015 Dec 24. PMID 26705192
- [Background] Baquerizo Nole KL, Yim E, Keri JE. Probiotics and prebiotics in dermatology. J Am Acad Dermatol. 2014 Oct;71(4):814-21. doi: 10.1016/j.jaad.2014.04.050. Epub 2014 Jun 4. PMID 24906613
- [Background] Costello EK, Lauber CL, Hamady M, Fierer N, Gordon JI, Knight R. Bacterial community variation in human body habitats across space and time. Science. 2009 Dec 18;326(5960):1694-7. doi: 10.1126/science.1177486. Epub 2009 Nov 5. PMID 19892944
- [Background] Dailey HA, Gerdes S, Dailey TA, Burch JS, Phillips JD. Noncanonical coproporphyrin-dependent bacterial heme biosynthesis pathway that does not use protoporphyrin. Proc Natl Acad Sci U S A. 2015 Feb 17;112(7):2210-5. doi: 10.1073/pnas.1416285112. Epub 2015 Feb 2. PMID 25646457
- [Background] Fitz-Gibbon S, Tomida S, Chiu BH, Nguyen L, Du C, Liu M, Elashoff D, Erfe MC, Loncaric A, Kim J, Modlin RL, Miller JF, Sodergren E, Craft N, Weinstock GM, Li H. Propionibacterium acnes strain populations in the human skin microbiome associated with acne. J Invest Dermatol. 2013 Sep;133(9):2152-60. doi: 10.1038/jid.2013.21. Epub 2013 Jan 21. PMID 23337890
- [Background] Gribbon EM, Cunliffe WJ, Holland KT. Interaction of Propionibacterium acnes with skin lipids in vitro. J Gen Microbiol. 1993 Aug;139(8):1745-51. doi: 10.1099/00221287-139-8-1745. PMID 8409917
- [Background] Johnson T, Kang D, Barnard E, Li H. Strain-Level Differences in Porphyrin Production and Regulation in Propionibacterium acnes Elucidate Disease Associations. mSphere. 2016 Feb 10;1(1):e00023-15. doi: 10.1128/mSphere.00023-15. eCollection 2016 Jan-Feb. PMID 27303708
- [Background] Kang D, Shi B, Erfe MC, Craft N, Li H. Vitamin B12 modulates the transcriptome of the skin microbiota in acne pathogenesis. Sci Transl Med. 2015 Jun 24;7(293):293ra103. doi: 10.1126/scitranslmed.aab2009. PMID 26109103
- [Background] Kasimatis G, Fitz-Gibbon S, Tomida S, Wong M, Li H. Analysis of complete genomes of Propionibacterium acnes reveals a novel plasmid and increased pseudogenes in an acne associated strain. Biomed Res Int. 2013;2013:918320. doi: 10.1155/2013/918320. Epub 2013 May 13. PMID 23762865
- [Background] Kishishita M, Ushijima T, Ozaki Y, Ito Y. New medium for isolating propionibacteria and its application to assay of normal flora of human facial skin. Appl Environ Microbiol. 1980 Dec;40(6):1100-5. doi: 10.1128/aem.40.6.1100-1105.1980. PMID 7470244
- [Background] Kjeldstad B, Johnsson A, Sandberg S. Influence of pH on porphyrin production in Propionibacterium acnes. Arch Dermatol Res. 1984;276(6):396-400. doi: 10.1007/BF00413361. PMID 6517611
- [Background] Kwon HH, Suh DH. Recent progress in the research about Propionibacterium acnes strain diversity and acne: pathogen or bystander? Int J Dermatol. 2016 Nov;55(11):1196-1204. doi: 10.1111/ijd.13282. PMID 27421121
- [Background] Lomholt HB, Kilian M. Population genetic analysis of Propionibacterium acnes identifies a subpopulation and epidemic clones associated with acne. PLoS One. 2010 Aug 19;5(8):e12277. doi: 10.1371/journal.pone.0012277. PMID 20808860
- [Background] McDowell A, Barnard E, Nagy I, Gao A, Tomida S, Li H, Eady A, Cove J, Nord CE, Patrick S. An expanded multilocus sequence typing scheme for propionibacterium acnes: investigation of 'pathogenic', 'commensal' and antibiotic resistant strains. PLoS One. 2012;7(7):e41480. doi: 10.1371/journal.pone.0041480. Epub 2012 Jul 30. PMID 22859988
- [Background] McDowell A, Nagy I, Magyari M, Barnard E, Patrick S. The opportunistic pathogen Propionibacterium acnes: insights into typing, human disease, clonal diversification and CAMP factor evolution. PLoS One. 2013 Sep 13;8(9):e70897. doi: 10.1371/journal.pone.0070897. eCollection 2013. PMID 24058439
- [Background] McDowell A, Perry AL, Lambert PA, Patrick S. A new phylogenetic group of Propionibacterium acnes. J Med Microbiol. 2008 Feb;57(Pt 2):218-224. doi: 10.1099/jmm.0.47489-0. PMID 18201989
- [Background] McGinley KJ, Webster GF, Ruggieri MR, Leyden JJ. Regional variations in density of cutaneous propionibacteria: correlation of Propionibacterium acnes populations with sebaceous secretion. J Clin Microbiol. 1980 Nov;12(5):672-5. doi: 10.1128/jcm.12.5.672-675.1980. PMID 7276142
- [Background] Meyer K, Pappas A, Dunn K, Cula GO, Seo I, Ruvolo E, Batchvarova N. Evaluation of Seasonal Changes in Facial Skin With and Without Acne. J Drugs Dermatol. 2015 Jun;14(6):593-601. PMID 26091385
- [Background] Mirshahpanah P, Maibach HI. Models in acnegenesis. Cutan Ocul Toxicol. 2007;26(3):195-202. doi: 10.1080/15569520701502815. PMID 17687685
- [Background] Nakatsuji T, Chen TH, Narala S, Chun KA, Two AM, Yun T, Shafiq F, Kotol PF, Bouslimani A, Melnik AV, Latif H, Kim JN, Lockhart A, Artis K, David G, Taylor P, Streib J, Dorrestein PC, Grier A, Gill SR, Zengler K, Hata TR, Leung DY, Gallo RL. Antimicrobials from human skin commensal bacteria protect against Staphylococcus aureus and are deficient in atopic dermatitis. Sci Transl Med. 2017 Feb 22;9(378):eaah4680. doi: 10.1126/scitranslmed.aah4680. PMID 28228596
- [Background] Sanchez A, Castro M, Castilla L, Guerrero P, Martin E. [Spontaneous peritonitis caused by Aeromonas hydrophila]. Enferm Infecc Microbiol Clin. 1989 Feb;7(2):112-3. No abstract available. Spanish. PMID 2490661
- [Background] Richter C, Trojahn C, Dobos G, Blume-Peytavi U, Kottner J. Follicular fluorescence quantity to characterize acne severity: a validation study. Skin Res Technol. 2016 Nov;22(4):451-459. doi: 10.1111/srt.12286. Epub 2016 Jan 25. PMID 26804729
- [Background] Shu M, Kuo S, Wang Y, Jiang Y, Liu YT, Gallo RL, Huang CM. Porphyrin metabolisms in human skin commensal Propionibacterium acnes bacteria: potential application to monitor human radiation risk. Curr Med Chem. 2013;20(4):562-8. doi: 10.2174/0929867311320040007. PMID 23231351
- [Background] Thiboutot D, Gollnick H, Bettoli V, Dreno B, Kang S, Leyden JJ, Shalita AR, Lozada VT, Berson D, Finlay A, Goh CL, Herane MI, Kaminsky A, Kubba R, Layton A, Miyachi Y, Perez M, Martin JP, Ramos-E-Silva M, See JA, Shear N, Wolf J Jr; Global Alliance to Improve Outcomes in Acne. New insights into the management of acne: an update from the Global Alliance to Improve Outcomes in Acne group. J Am Acad Dermatol. 2009 May;60(5 Suppl):S1-50. doi: 10.1016/j.jaad.2009.01.019. PMID 19376456
- [Background] Tomida S, Nguyen L, Chiu BH, Liu J, Sodergren E, Weinstock GM, Li H. Pan-genome and comparative genome analyses of propionibacterium acnes reveal its genomic diversity in the healthy and diseased human skin microbiome. mBio. 2013 Apr 30;4(3):e00003-13. doi: 10.1128/mBio.00003-13. PMID 23631911
- [Background] Walsh TR, Efthimiou J, Dreno B. Systematic review of antibiotic resistance in acne: an increasing topical and oral threat. Lancet Infect Dis. 2016 Mar;16(3):e23-33. doi: 10.1016/S1473-3099(15)00527-7. Epub 2016 Feb 5. PMID 26852728
- [Background] Wei EX, Kirsner RS, Eaglstein WH. End points in dermatologic clinical trials: A review for clinicians. J Am Acad Dermatol. 2016 Jul;75(1):203-9. doi: 10.1016/j.jaad.2016.01.052. Epub 2016 Feb 28. PMID 26936300
- See also: [ClinicalTrials.gov] Investigator Assessment Tolerability Scoring: A Study to Evaluate Tolerability of Two Topical Drug Products in the Treatment of Facial Acne. Received: August 2009; Updated: October 2016. — http://clinicaltrials.gov/ct2/show/NCT00964223
- See also: DermNet New Zealand. Acne vulgaris: Acne Grading — http://www.dermnetnz.org/topics/acne-vulgaris
- See also: [FDA] Guidance for Industry: Acne Vulgaris: Developing Drugs for Treatment. Draft: September 2005 — http://www.fda.gov/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM071292
- See also: Investigator Assessment Tolerability Scoring. A Study to Evaluate Tolerability of Two Topical Drug Products in the Treatment of Facial Acne, 2009; updated 2016 — http://clinicaltrials.gov/ct2/show/study/NCT00964223
- See also: Propionibacterium acnes e a resistência bacteriana [Propionibacterium acnes and bacterial resistance] — http://www.surgicalcosmetic.org.br/detalhe-artigo/404
- See also: Propionibacteriales ord. Nov. In: Whitman W, et al. eds. Bergey's Manual of Systematic Bacteriology — http://www.springer.com/us/book/9780387950433

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose: 10^4 CFU/cm^2 NB01 colony forming unit (CFU)
- High Dose: 10^5 CFU/cm^2 NB01 colony forming unit (CFU)
Period: Overall Study
Arm/Group | Low Dose | High Dose
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Dose: 10^4 CFU/cm^2 NB01
- High Dose: 10^5 CFU/cm^2 NB01
- Total: Total of all reporting groups
Arm/Group | Low Dose | High Dose | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.6 (4.77) | 26.6 (3.78) | 24.6 (4.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 4 | 2 | 6
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Reproductive Status [Count of Participants; unit: Participants]
  Able to bear children | 5 | 4 | 9
  Total abstinence (male) | 0 | 1 | 1
Method of Contraception (Female) [Count of Participants; unit: Participants] — Note only females in Low Dose, one male in High Dose.
  Participants
    Total abstinence | 2 | 0 | 2
    Barrier method with spermicide | 3 | 0 | 3
    Oral, injected or implanted combined hormonal meth | 0 | 4 | 4
    male subject: not recorded | 0 | 1 | 1
Investigator's Global Assessment (IGA) Score - Face [Mean (Standard Deviation); unit: units on a scale] — The investigator assessed the participant's inflammatory lesions on the face using the IGA 5-point scale at screening visit.
  The scale ranges from 0 (best): clear, to 4 (worst).
  units on a scale | 3 (0) | 3 (0) | 3 (0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Engraftment of Probiotic Following a Single Application.
Description: Engraftment is defined as the percentage of bacteria recovered from hair follicles that are health-associated (NB01) as measured with proprietary quantitative polymerase chain assays. Successful follicular engraftment, defined as both deoR/PanBac >40% and Cas5/PanBac >40% in the Day 2 (24H) ) Biore Strip samples. Cas5/PanBac and deoR/PanBac are the percentages of bacteria in a sample containing the CRISPR associated protein Cas5 and a repressor of porphyrin production deoR, respectively. Pan-Bacterial (PanBac) is a loci found in nearly all bacteria found on the face and thus serves as the denominator to calculate the percentage of bacteria with any loci.
Time Frame: 2 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 5 | 5
Participants | 2 | 1

2. Primary Outcome: Dose Schedule Determination Based on Time to Peak deoR and Cas5
Description: To determine longevity of the live biotherapeutic after a single application, swab samples were collected at Baseline, 6, 24 and 48 hours after application, and genotyped as above. For each participant the absolute change, from Baseline, in the percentage of the two loci present in the live biotherapeutic (deoR and Cas5) were calculated. A significant positive change is indicative of the continued presence of the live biotherapeutic.
Time Frame: From Baseline to 48 hours after application
Measure: Mean (Standard Deviation); unit: % of total bacteria w/ genotype
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 5 | 5
% of total bacteria w/ genotype
  Genotype 1 (deoR), 6 hours | -0.4 (36.3) | 51.2 (28.6)
  Genotype 1 (deoR), 24 hours | -4.2 (25.7) | 5.2 (7.6)
  Genotype 1 (deoR), 48 hours | 13.8 (33.5) | 2.8 (10.9)
  Genotype 2 (Cas 5), 6 hours | 12.8 (27.9) | 48.4 (21.7)
  Genotype 2 (Cas 5), 24 hours | 3.4 (15.6) | 4.4 (8.8)
  Genotype 2 (Cas 5), 48 hours | 3.2 (12.2) | 1.8 (12.1)

3. Primary Outcome: Number of Participants With Change in Investigator Global Assessment (IGA) Score
Description: Number of participants with a changed Investigator Global Assessment (IGA) score after single application of NB01; positive number if grade is reduced (e.g. from 3 to 2) or negative number is IGA grade increased.
  The Investigator Global Assessment 5-Point Score is a standard FDA acne assessment tool with scoring as follows:
  Grade 0-Clear (Clear skin with no inflammatory or non-inflammatory lesions. The category of clear should represent true absence of disease) Grade1-Almost Clear (A few scattered comedones and no more than one small papule) Grade 2-Mild (Some comedones, some papules and pustules; no nodules) Grade 3-Moderate (Many comedones, papules and pustules; one nodule may be present) Grade 4-Severe (Covered with comedones, numerous papules and pustules and no more than a few nodular lesions)
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 5 | 5
Participants
  Participants with changed IGA @ 6 hours | 0 | 0
  Participants with changed IGA @ 1 day | 0 | 0
  Participants with changed IGA @ 2 days | 0 | 0
  Participants with changed IGA @ 6 days | 0 | 0
  Participants with changed IGA @ 28 days | 2 | 0

4. Primary Outcome: Safety Profile and Tolerability of a Singly Applied NB01 Using Acne Lesion Counts.
Description: Absolute Lesion Count: All Lesions for the Whole Face; with higher numbers of lesion representing worsening or more severe acne
Time Frame: From Screening to 28 days after application, typically 2 months
Population: All participants who received at least one dose of treatment.
Measure: Mean (Standard Deviation); unit: count of lesions
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 5 | 5
count of lesions
  Screening | 49.4 (21.08) | 38.8 (16.60)
  Day 1 (0 hours) | 22.6 (13.26) | 42.6 (3.8)
  Day 1 (6 hours) | 21.0 (9.22) | 39.8 (25.41)
  Day 2 | 31.6 (3.51) | 38.2 (25.29)
  Day 3 | 32.2 (6.18) | 35.4 (24.17)
  Day 7 | 25.6 (4.72) | 34.2 (19.11)
  Day 28 | 25.8 (14.31) | 32.6 (59.22)

5. Primary Outcome: Number of Participants With Change in Investigator Assessment of Tolerability Score: Skin Peeling
Description: Safety profile and tolerability of a singly applied NB01 using the Investigator Assessment of Tolerability Scoring (0 = None; 1 = Slight; 2 = Moderate; 3 = Intense) for Skin Peeling. Reference: ClinicalTrials.gov: Investigator Assessment Tolerability Scoring: A Study to Evaluate Tolerability of Two Topical Drug Products in the Treatment of Acne.
Time Frame: From Screening to 28 days after application, typically 2 months
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 5 | 5
Participants
  Screening, scale = 0 (none) | 3 | 5
  Screening, scale = 1 (slight) | 2 | 0
  Day 1 (0 hours), scale = 0 (none) | 4 | 5
  Day 1 (0 hours), scale = 1 (slight) | 1 | 0
  Day 1 (6 hours), scale = 0 (none) | 4 | 5
  Day 1 (6 hours), scale = 1 (slight) | 1 | 0
  Day 2, scale = 0 (none) | 5 | 5
  Day 3, scale = 0 (none) | 5 | 5
  Day 7, scale = 0 (none) | 5 | 5
  Day 28, scale = 0 (none) | 5 | 5

6. Primary Outcome: Number of Participants With Change in Investigator Assessment of Tolerability Score: Irritant/Allergic Contact Dermatitis
Description: Safety profile and tolerability of a singly applied NB01 using the Investigator Assessment of Tolerability Scoring (0 = None; 1 = Slight; 2 = Moderate; 3 = Intense) for Irritant/Allergic Contact Dermatitis. Reference: ClinicalTrials.gov: Investigator Assessment Tolerability Scoring: A Study to Evaluate Tolerability of Two Topical Drug Products in the Treatment of Acne.
Time Frame: From Screening to 28 days after application, typically 2 months
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 5 | 5
Participants
  Screening, scale = 0 (none) | 5 | 5
  Day 1 (0 hours), scale = 0 (none) | 5 | 5
  Day 1 (6 hours), scale = 0 (none) | 5 | 5
  Day 2, scale = 0 (none) | 5 | 5
  Day 3, scale = 0 (none) | 5 | 5
  Day 7, scale = 0 (none) | 5 | 5
  Day 28, scale = 0 (none) | 5 | 5

7. Primary Outcome: Number of Participants With Change in Investigator Assessment of Tolerability Score: Hyperpigmentation
Description: Safety profile and tolerability of a singly applied NB01 using the Investigator Assessment of Tolerability Scoring (0 = None; 1 = Slight; 2 = Moderate; 3 = Intense) for Hyperpigmentation. Reference: ClinicalTrials.gov: Investigator Assessment Tolerability Scoring: A Study to Evaluate Tolerability of Two Topical Drug Products in the Treatment of Acne.
Time Frame: From Screening to 28 days after application, typically 2 months
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 5 | 5
Participants
  Screening, scale = 0 (none) | 5 | 5
  Day 1 (0 hours), scale = 0 (none) | 5 | 5
  Day 1 (6 hours), scale = 0 (none) | 5 | 5
  Day 2, scale = 0 (none) | 5 | 5
  Day 3, scale = 0 (none) | 5 | 5
  Day 7, scale = 0 (none) | 5 | 5
  Day 28, scale = 0 (none) | 5 | 5

8. Primary Outcome: Number of Participants With Change in Investigator Assessment of Tolerability Score: Ocular Irritation
Description: Safety profile and tolerability of a singly applied NB01 using the Investigator Assessment of Tolerability Scoring (0 = None; 1 = Slight; 2 = Moderate; 3 = Intense) for Ocular Irritation. Reference: ClinicalTrials.gov: Investigator Assessment Tolerability Scoring: A Study to Evaluate Tolerability of Two Topical Drug Products in the Treatment of Acne.
Time Frame: From Screening to 28 days after application, typically 2 months
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 5 | 5
Participants
  Screening, scale = 0 (none) | 5 | 5
  Day 1 (0 hours), scale = 0 (none) | 5 | 5
  Day 1 (6 hours), scale = 0 (none) | 5 | 5
  Day 2, scale = 0 (none) | 5 | 5
  Day 3, scale = 0 (none) | 5 | 5
  Day 7, scale = 0 (none) | 5 | 5
  Day 28, scale = 0 (none) | 5 | 5

9. Primary Outcome: Number of Participants With Change in Investigator Assessment of Tolerability Score: Conjunctival Injection
Description: Safety profile and tolerability of a singly applied NB01 using the Investigator Assessment of Tolerability Scoring (0 = None; 1 = Slight; 2 = Moderate; 3 = Intense) for Conjunctival Injection. Reference: ClinicalTrials.gov: Investigator Assessment Tolerability Scoring: A Study to Evaluate Tolerability of Two Topical Drug Products in the Treatment of Acne.
Time Frame: From Screening to 28 days after application, typically 2 months
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 5 | 5
Participants
  Screening, scale = 0 (none) | 5 | 5
  Day 1 (0 hours), scale = 0 (none) | 5 | 5
  Day 1 (6 hours), scale = 0 (none) | 5 | 5
  Day 2, scale = 0 (none) | 5 | 5
  Day 3, scale = 0 (none) | 5 | 5
  Day 7, scale = 0 (none) | 5 | 5
  Day 28, scale = 0 (none) | 5 | 5

10. Primary Outcome: Number of Participants With Change in Investigator Assessment of Tolerability Score: Mucosal Toxicity
Description: Safety profile and tolerability of a singly applied NB01 using the Investigator Assessment of Tolerability Scoring (0 = None; 1 = Slight; 2 = Moderate; 3 = Intense) for Mucosal Toxicity. Reference: ClinicalTrials.gov: Investigator Assessment Tolerability Scoring: A Study to Evaluate Tolerability of Two Topical Drug Products in the Treatment of Acne.
Time Frame: From Screening to 28 days after application, typically 2 months
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 5 | 5
Participants
  Screening, scale = 0 (none) | 5 | 5
  Day 1 (0 hours), scale = 0 (none) | 5 | 5
  Day 1 (6 hours), scale = 0 (none) | 5 | 5
  Day 2, scale = 0 (none) | 5 | 5
  Day 3, scale = 0 (none) | 5 | 5
  Day 7, scale = 0 (none) | 5 | 5
  Day 28, scale = 0 (none) | 5 | 5

11. Primary Outcome: Number of Participants With Change in Investigator Assessment of Tolerability Score: Skin Erythema.
Description: Safety profile and tolerability of a singly applied NB01 using the Investigator Assessment of Tolerability Scoring (0 = None; 1 = Slight; 2 = Moderate; 3 = Intense) for Skin Erythema. Reference: ClinicalTrials.gov: Investigator Assessment Tolerability Scoring: A Study to Evaluate Tolerability of Two Topical Drug Products in the Treatment of Acne.
Time Frame: From Screening to 28 days after application, typically 2 months
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 5 | 5
Participants
  Screening, scale = 0 (none) | 2 | 5
  Screening, scale = 1 (slight) | 3 | 0
  Day 1 (0 hours), scale = 0 (none) | 3 | 5
  Day 1 (0 hours), scale = 1 (slight) | 1 | 0
  Day 1 (0 hours), scale = 2 (moderate) | 1 | 0
  Day 1 (6 hours), scale = 0 (none) | 3 | 5
  Day 1 (6 hours), scale = 1 (slight) | 1 | 0
  Day 1 (6 hours), scale = 2 (moderate) | 1 | 0
  Day 2, scale = 0 (none) | 4 | 5
  Day 2, scale = 1 (slight) | 1 | 0
  Day 3, scale = 0 (none) | 4 | 5
  Day 3, scale = 1 (slight) | 1 | 0
  Day 7, scale = 0 (none) | 4 | 5
  Day 7, scale = 1 (slight) | 1 | 0
  Day 28, scale = 0 (none) | 5 | 5

12. Primary Outcome: Number of Participants With Change in Investigator Assessment of Tolerability Score: Skin Dryness.
Description: Safety profile and tolerability of a singly applied NB01 using the Investigator Assessment of Tolerability Scoring (0 = None; 1 = Slight; 2 = Moderate; 3 = Intense) for Skin Dryness. Reference: ClinicalTrials.gov: Investigator Assessment Tolerability Scoring: A Study to Evaluate Tolerability of Two Topical Drug Products in the Treatment of Acne.
Time Frame: From Screening to 28 days after application, typically 2 months
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 5 | 5
Participants
  Screening, scale = 0 (none) | 4 | 5
  Screening, scale = 1 (slight) | 1 | 0
  Day 1 (0 hours), scale = 0 (none) | 4 | 5
  Day 1 (0 hours), scale = 1 (slight) | 1 | 0
  Day 1 (6 hours), scale = 0 (none) | 4 | 5
  Day 1 (6 hours), scale = 1 (slight) | 1 | 0
  Day 2, scale = 0 (none) | 4 | 5
  Day 2, scale = 1 (slight) | 1 | 0
  Day 3, scale = 0 (none) | 4 | 5
  Day 3, scale = 1 (slight) | 1 | 0
  Day 7, scale = 0 (none) | 5 | 5
  Day 28, scale = 0 (none) | 3 | 5
  Day 28, scale = 1 (slight) | 2 | 0

ADVERSE EVENTS:
Time Frame: From Screening to 28 days after application, typically 2 months
Arm/Group | Low Dose | High Dose
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/5 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=5) | High Dose (N=5)
Application site dermatitis (General disorders) | 1 (1) | 0 (0) — ADMINISTRATION SITE CONDITIONS
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/69/NCT03450369/Prot_SAP_000.pdf